CLINICAL TRIAL: NCT06562270
Title: CorEvitas International Adolescent Alopecia Areata (AA) Drug Safety and Effectiveness Registry
Status: Recruiting | Type: Observational
Sponsor: CorEvitas (Network)
Responsible Party: Sponsor
Other Study IDs: CorEvitas-AA-565
Record Dates: First submitted 2024-07-30; First posted 2024-08-20 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective observational registry focusing on an adolescent cohort diagnosed with severe alopecia areata,receiving routine care from dermatology providers. Visit schedules for patients will be determined by the provider in accordance with routine clinical care, and any prescriptions provided to patients will adhere to product availability and local prescribing guidelines/regulations in the country where the participating registry site is located.

DETAILED DESCRIPTION:
The objective of the registry is to create a cohort of adolescent subjects to evaluate the long-term real-world safety and effectiveness of routine clinical care of treatments for severe AA. Data collected through the registry may be used to address a range of research questions and use cases including, but not limited to: better characterizing the natural history of the disease, evaluating the effectiveness and safety of commercially available medications for the treatment of severe AA in adolescents, providing information to support characterization of adolescent growth and development and ongoing risk-benefit evaluation by drug manufacturers and regulators, and research related to drug utilization, disease burden, and unmet needs. Further, data collected may be used to generate real world evidence to inform clinical decision making by patients and treating providers.

This will be enabled through standardized data collection including validated instruments for patient-reported outcomes (PROs) and clinician-reported outcomes (ClinROs), the active evaluation of prevalent and incident comorbidities and adverse events, and the recording of medication utilization data.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in this registry, an individual must meet all the following criteria:

1. Has ever been diagnosed with severe AA by a dermatologist or a qualified dermatology provider.
2. Is 12-17 years of age at the time of enrollment.
3. Is willing to provide consent/assent for participation in the registry.
4. Has been prescribed a new commercially available advanced therapy and/or conventional systemic therapy for the treatment of severe AA in adolescents in the context of routine clinical care that is consistent with local prescribing guidelines and/or regulations for the country where the site is located.

A new therapy is a medication that the subject has never taken before.

1. At the time of registry enrollment OR
2. Within 6 months prior to registry enrollment In the opinion of the treating provider, is deemed a candidate for treatment with a commercially available advanced therapy and/or conventional systemic therapy for the treatment of severe AA in adolescents but has not received nor is planning to initiate treatment at the time of registry enrollment.

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in the registry:

1. Is participating or planning to participate in a blinded clinical trial for any investigational medication.
2. Is unwilling or unable to provide standing height measurements.

Ages: 12 Years to 17 Years | Sex: All
Age Groups: Child
Study Population: Subjects can enroll as early as age 12 and will be followed until the age of 18; therefore, the maximum duration a subject can be enrolled is 6 years.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2024-03-07 (Actual); Primary Completion 2099-12-31 (Estimated); Study Completion 2099-12-31 (Estimated)

PRIMARY OUTCOMES:
AA epidemiology, presentation, natural history, management, and outcomes | Through Study completion until the subject is 18 years
  The major clinical outcomes include an assessment of the epidemiology of Alopecia Areata; to better understand the presentation, natural history, management and outcomes.

SECONDARY OUTCOMES:
Percentage of patients with history of comorbidities | at registry enrollment
  Data collected through the registry may be used to address a range of research questions and use cases including, but not limited to: better characterizing the natural history of the disease, evaluating the effectiveness and safety of commercially available medications for the treatment of severe AA in adolescents, providing information to support characterization of adolescent growth and development and ongoing risk-benefit evaluation by drug manufacturers and regulators, and research related to drug utilization, disease burden, and unmet needs
Patient reported : Hair Concealment Question | every 6 months until the subject is 18 years
  Helps to determine alopecia
Patient reported : Stressful Life Event | every 6 months until the subject is 18 years
  Determines correlation between the disease & stressful life events
Patient reported : Scalp Hair Assessment | every 6 months until the subject is 18 years
  Determines hair loss
Patient reported :Measures for Eye Irritation & Nail Appearance | every 6 months until the subject is 18 years
  Determines eye irritation & nail appearance due to alopecia
Patient reported : Numerical Rating Scale for Nasal irritation | every 6 months until the subject is 18 years
  Determines nasal irritation due to alopecia
Patient reported : Alopecia Areata Patient Priority Outcomes (AAPPO) | every 6 months until the subject is 18 years
  To assess the consequences associated with Alopecia Areata (AA) of the highest priority to the patients, including hair loss signs, emotional symptoms, and activity limitations
Patient reported : Patient Health Questionnaire (PHQ) | every 6 months until the subject is 18 years
  Determines depression in subjects with alopecia
Patient reported :PROMIS Pediatric Sleep Disturbance 4 a | every 6 months until the subject is 18 years
  Determines sleep disturbance in subjects with alopecia
Patient reported : PROMIS Pediatric Stigma 8a | every 6 months until the subject is 18 years
  Determines Stigma in subjects with alopecia
Patient reported : Grief Assessment | every 6 months until the subject is 18 years
  Determines level of grief in subjects with alopecia
Patient reported : Pubertal Tanner Staging | every 6 months until the subject is 18 years
  Determines pubertal progression
Physician reported : Pubertal Progression: Tanner Staging Assessment | Every six Months until a subject is 18 years or the subjects reaches stage 5 of the tanner stangings assessment
  Determines pubertal progression
Physician reported : Severity of Alopecia Tool (SALT) | every 6 months until the subject is 18 years
  Determines percentage for hair loss & ranges from 0 to 100
Physician reported : Alopecia Areata Investigator Global Assessment Scale (AA-IGA) | every 6 months until the subject is 18 years
  Helps in clinical evaluation of Alopecia Aareata
Physician reported : Measures for Eyebrow & Eyelash Hair loss and Nail Appearance | every 6 months until the subject is 18 years
  Determines hair loss in patients with alopecia aareata

CONTACTS AND LOCATIONS:
Locations (1):
- CorEvitas, LLC, Waltham, Massachusetts, United States